CLINICAL TRIAL: NCT05791851
Title: Heplisav-B Revaccination for Hepatitis B Vaccine Nonresponders
Acronym: HBR2
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Baltimore VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Meagan Deming, Assistant Professor, University of Maryland, Baltimore
Other Study IDs: HP-83378
Record Dates: First submitted 2023-03-07; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: HIV Infections; Hepatitis B; Vaccine Response Impaired
Keywords: Heplisav-B; HIV; vaccine
MeSH Terms: conditions — HIV Infections; Hepatitis B

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HIV infected
- HIV uninfected

SUMMARY:
The goal of this natural history study is to examine the immune responses to the Heplisav-B vaccine in Veterans living with HIV who were non-responders to prior HBV vaccination. A comparison group of HBV vaccine nonresponders without HIV infection will be enrolled to characterize the HIV-associated immune alterations that affect vaccine response. The investigators hypothesize that TLR9-mediated innate immune stimulation with Heplisav will elicit HBV seroprotection despite prior vaccination failures in persons living with HIV, compared to HIV uninfected individuals.

Participants eligible for Heplisav-B vaccination will be asked to provide blood samples at multiple timepoints before and after their vaccination.

DETAILED DESCRIPTION:
HIV-positive individuals are at increased risk of morbidity and mortality from Hepatitis B co-infection, due to shared routes of transmission, increased likelihood of developing chronic infection (as opposed to spontaneous clearance), and increased immune dysregulation leading to accelerated disease progression, and so current guidelines recommend the routine vaccination of HIV-positive individuals against HBV. However, because achieved seroprotection rates (SPR) are historically lower than in HIV-negative individuals, post-vaccination serologic testing is recommended for this group and re-vaccination (with increased dose or additional doses) should be attempted for those who were non-responders to the initial vaccine. Heplisav-B is a HBV vaccine adjuvanted with a TLR9 agonist that has shown improved SPR among groups with reduced response rates to classic alum-adjuvanted vaccines, such as those with CKD, obesity, or diabetes. The investigators propose to evaluate immunological mechanisms of protection in Veterans who were non-responders to prior HBV vaccination now receiving Heplisav vaccinations. The investigators will enroll a comparison group of HIV-negative individuals to characterize the HIV-associated immune alterations that modulate vaccine response. The investigators hypothesize that TLR9-mediated innate immune stimulation with Heplisav will elicit HBV seroprotection despite prior vaccination failures in persons living with HIV, compared to HIV uninfected individuals. By assessing innate immune responses and B cell immunophenotypes at baseline, post-vaccination, and at long-term followup in Veterans with and without HIV the investigators will assess the mechanisms by which the immunostimulatory effects of TLR9 agonists may overcome the immune dysfunction in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 by age of screening
* If HIV positive, either:

  * Suppressed on a stable, ARV regimen for >4 weeks with CD4 count >100. HIV VL suppressed <50 copies/mL, although single isolated VL >50 not excluded.

OR

* Untreated ≥ 8 weeks with CD4 count >100

  * Prior HBV vaccine (other than Heplisav) with last dose >30 days prior to screening and anti-HBSAg ≤10 IU/mL measured >30days from last vaccine dose. (No exclusion for HBV CAb positive.)
  * Ability to provide informed consent and adhere to clinic visits (in the judgment of both the participant and the provider)
  * No history of adverse reaction to HBV vaccines or components thereof
  * If HCV Ab positive: undetectable HCV viral load and >12 weeks from completion of any HCV therapy.

Exclusion Criteria:

* History of allergic reaction to HBV vaccines or components (including yeast)
* HBsAb titer >10 IU/mL on screening evaluation
* Clinically significant illness (other than HIV) that may, in the opinion of the investigator, interfere with the subject treatment, or adherence to protocol. This may include but is not limited to a history of transplant, decompensated cirrhosis, or malignancy that may interfere with host immunity.
* Poor venous access interfering with blood sample collection
* Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.
* No exclusion will be made for chronic renal disease or ESRD

Ages: 18 Years to 109 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population includes patients (or healthcare providers) who have received prior Hepatitis B vaccines without achieving seroprotection (defined as a negative SAb qualitative titer or a SAb quantitative titer <10 mIU/mL collected at least 30 days after last vaccine dose). The primary enrollment group will include Veterans living with HIV, with a comparator group of HIV-negative individuals. An additional exploratory population of HBV vaccine nonresponders who were successfully treated for HCV infection may be included to provide an opportunity for evaluation of the immune responses in patients who have been cured of chronic viral infections.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Change in B cell functional responses | Day 30
  Characterize the change in B cell functional responses by ELISpot on day 30 compared to baseline
Change in B cell functional responses | Day 60
  Characterize the change in B cell functional responses by ELISpot on day 60 compared to baseline
Change in B cell functional responses | Day 365
  Characterize the change in B cell functional responses by ELISpot on day 365 compared to baseline
Change in B cell phenotypic responses | Day 30
  Characterize the change in B cell phenotypic responses by flow cytometry on day 365 compared to baseline
Change in B cell phenotypic responses | Day 60
  Characterize the change in B cell phenotypic responses by flow cytometry on day 365 compared to baseline
Change in B cell phenotypic responses | Day 365
  Characterize the change in B cell phenotypic responses by flow cytometry on day 365 compared to baseline
Cytokine profile | Day 1
  Change in cytokine profile on day 1 compared to baseline

SECONDARY OUTCOMES:
Hepatitis B surface antibody responses | Day 30
  Characterization of the hepatitis B surface antibody titers on day 30 compared to baseline
Hepatitis B surface antibody responses | Day 60
  Characterization of the hepatitis B surface antibody titers on day 60 compared to baseline
Hepatitis B surface antibody responses | Day 365
  Characterization of the hepatitis B surface antibody titers on day 365 compared to baseline
Hepatitis B surface antibody response rates | Day 30
  Characterization of the hepatitis B surface antibody response rates on day 30 compared to baseline
Hepatitis B surface antibody response rates | Day 60
  Characterization of the hepatitis B surface antibody response rates on day 60 compared to baseline
Hepatitis B surface antibody response rates | Day 365
  Characterization of the hepatitis B surface antibody response rates on day 365 compared to baseline

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Baltimore Veterans Affairs Medical Center, Baltimore, Maryland
  - Institute of Human Virology, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No